CLINICAL TRIAL: NCT05869656
Title: THIRST Alert Trial - a Randomised Controlled Trial Within the Electronic Health Record of an Interruptive Alert Displaying a Fluid Restriction Suggestion in Patients With the Treatable Trait of Congestion
Brief Title: THIRST Alert Trial
Acronym: THIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (UCLH) NHS Foundation Trust (Unknown); National Institute for Health and Care Research (NIHR) UCLH Biomedical Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 151938
Record Dates: First submitted 2023-04-26; First posted 2023-05-22 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Fluid Overload; Congestive Heart Failure
Keywords: Electronic health record; Comparative effectiveness research; Pragmatic trial; Learning health systems; Heart Failure; Treatable trait
MeSH Terms: conditions — Edema; Heart Failure

STUDY DESIGN:
Intervention Model Description: Feasibility RCT with an alert intervention that is clinician facing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alert recommending oral fluid restriction (Experimental): The alert will suggest to the treating clinician to fluid restrict the patient to 1L of oral fluid per day
  Interventions: Behavioral: Fluid restriction
- Alert recommending no oral fluid restriction (Active Comparator): The alert will suggest to the treating clinician to continue without any oral fluid restriction
  Interventions: Behavioral: Free fluids

INTERVENTIONS:
Behavioral: Fluid restriction — Oral fluid restriction of 1000ml per day
  Arms: Alert recommending oral fluid restriction
Behavioral: Free fluids — Continue care without any oral fluid restriction
  Arms: Alert recommending no oral fluid restriction

SUMMARY:
The aim of this feasibility study is to determine whether an alert embedded within the electronic health record (EHR) causes clinicians to enrol patients into a randomised controlled trial (RCT) comparing oral fluid restriction versus no restriction in patients admitted to hospital with fluid overload.

One of the main causes of fluid overload is heart failure where there is a lack of strong evidence to support the effectiveness of oral fluid restriction in the acute setting. This causes significant variation in clinical practice where decisions on whether or not to impose a restriction in oral fluid intake is based on the preference of the treating clinician rather than robust evidence from research.

THIRST Alert is a pragmatic randomised controlled trial (RCT), embedded in the EHR, which seeks to determine whether a computerised alert for the clinical team can change clinician behaviour during routine NHS care at University College London Hospitals NHS Foundation Trust (UCLH).

Patients with suspected fluid overload will be identified based on the prescription of intravenous furosemide, a medication used to stimulate diuresis (increased urine output) to remove excess fluid. A repeat prescription of intravenous furosemide within the first 48 hours of an unplanned admission will trigger the alert.

A clinician from the treating team will then be asked to consider enrolling the patient into the RCT if they judge that oral fluid restriction might be beneficial but they have uncertainty about this (clinical equipoise). Enrolled patients will be randomised to either oral fluid restriction of 1 litre per day or no fluid restriction. This will then be actioned through documenting as part of the clinical plan in the patients record and then communicated to the patient and the rest of the clinical team, including nursing staff.

The study will record the number of patients recruited into the trial and the effect of the alert on enrolled patients' subsequent oral fluid intake. There are no additional tests or follow up for patients and the trial finishes on discharge from the study site. All trial outcomes will use data collected from routine care and the study is supported by the UCLH Biomedical Research Centre, funded by NIHR.

DETAILED DESCRIPTION:
Trial Design:

A single centre, pragmatic, parallel group randomised controlled trial and feasibility study. The study will be conducted entirely within University College Hospital, at University College London Hospitals NHS Foundation Trust.

Research Hypothesis:

Clinician-facing alerts, delivered through the electronic health records system, provide a feasible method of enrolling patients into pragmatic trials evaluating the effectiveness of routine treatments

Clinical Research question:

In hospitalised patients with fluid overload, does an automated clinician-facing computerised decision support system (CDSS) alert recommendation for either oral fluid restriction (to 1L per day) or no-fluid restriction (continue with free fluids) result in a change in clinical behaviour and change in the oral fluid intake of enrolled patients?

Study participants:

The study population will be patients treated for suspected fluid overload with a regular prescription of intravenous (IV) furosemide within 48 hours of an unplanned hospital admission.

For staff participants, any clinician with prescribing rights for IV furosemide may be exposed to the CDSS alert. For subsequent medical staff, nursing staff and other allied health professionals, patient enrolment into the trial and their treatment allocation status will be communicated through both EHR and clinical processes that are embedded within routine care, including verbal and non-digital patient handover.

Summary of Interventions:

This study will evaluate the effect of a Best practice advisory (BPA) interruptive alert that is embedded within the electronic health record (EHR) used at the study site. The first BPA will ask the treating clinician whether they judge randomisation to either oral fluid restriction or no restriction is appropriate - if yes is selected, randomised allocation to one of two subsequent alerts will occur at the point of care. This intervention will be tested in silico prior to deployment to the live EHR.

Ethics:

This study protocol was approved by the London Riverside Research Ethics Committee (Ref: 22/LO/0889) and sponsored by University College London (Ref: 151938).

ELIGIBILITY:
Inclusion Criteria:

* Prescribed IV furosemide during the first 48h of their admission as a regular prescription rather than a one-off dose.
* Assessed as being suitable for inclusion in the trial by the responsible clinical team i.e., fluid restriction deemed to be in equipoise.

Exclusion Criteria:

* On a surgical, obstetric or critical care ward environment
* Patients who opt out of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited into the trial | 3 months
  The number of patients in which the usual care team thought there was equipoise for oral fluid restriction
Difference in oral fluid intake between intervention and control arms | 48 hours after randomisation
  Difference in documented oral intake (ml)

SECONDARY OUTCOMES:
Adherence to randomised alert recommendation | During trial recruitment window (up to day 2)
  Proportion of alerts actioned with corresponding clinical documentation
Proportion of alerts with clinical orders for nursing staff | During trial recruitment window (up to day 2)
  Corresponding documentation of nursing receipt of treatment allocation
Oral fluid intake | From date of randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  Documented oral fluid intake (ml)
Net fluid balance | From date of randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  Documented overall fluid balance (ml)
Weight change after randomisation | 48 hours after randomisation
  Weight (kg)
Length of stay | From day of admission to day of discharge, assessed up to 120 days after trial start date
  Number of Days
Frequency of blood test measurements of renal function | From date of randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  Number of times blood tests are measured
Prescription of Diuretic medications | From date of randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  Dose and duration of intravenous and oral diuretics
Daily change in creatinine | From 48 hours after randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  48 hours after randomisation
Patient reported outcome measure | From date of randomisation until date of hospital discharge, assessed up to 120 days after trial start date
  Visual analog scale (1-10) of wellbeing, thirst perception and breathlessness

CONTACTS AND LOCATIONS:
Overall Officials: Yang Chen, BMBCh, MSc, Principal Investigator — UCL; Tom Lumbers, MBBChir, PhD, Study Chair — UCL; Anoop D Shah, MBBS, PhD, Principal Investigator — UCL
Locations (1):
- University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Shah A, Jani Y, Higgins D, Saleem N, Chafer K, Sydes MR, Asselbergs FW, Lumbers RT. Rationale and design of the THIRST Alert feasibility study: a pragmatic, single-centre, parallel-group randomised controlled trial of an interruptive alert for oral fluid restriction in patients treated with intravenous furosemide. BMJ Open. 2024 Jan 11;14(1):e080410. doi: 10.1136/bmjopen-2023-080410. PMID 38216198